CLINICAL TRIAL: NCT03161574
Title: FOLFOXIRI Chemotherapy Alone as Neoadjuvant Treatment for MRI-defined Circumferential Radial Margin (CRM) Positive Rectal Cancer
Brief Title: FOLFOXIRI Chemotherapy Alone as Neoadjuvant Treatment for Circumferential Radial Margin (CRM) Positive Rectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants were recruited
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Wu Liucheng, Attending Physician, Guangxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FOLOXIRIREC
Record Dates: First submitted 2017-05-18; First posted 2017-05-22 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Rectal Cancer
Keywords: neochemotherapy; CRM
MeSH Terms: conditions — Rectal Neoplasms | interventions — FOLFOXIRI protocol; Fluorouracil; Oxaliplatin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FOLFOXIRI (Experimental): patients with CRM positive who received FOLFOXIRI alone for 6 cycles before surgery
  Interventions: Drug: FOLFOXIRI

INTERVENTIONS:
Drug: FOLFOXIRI — irinotecan* 165 mg/m² + oxaliplatin 85 mg/m² + leucovorin 200 mg/m² + 5FU 2800 mg/m² cont. inf. 46h all on day 1 of each 2 weeks cycle
  Other Names: 5-Fluorouracil; Oxaliplatin; Irinotecan

SUMMARY:
Neoadjuvant 5-Fu based chemoradiation followed by surgery is a standard treatment for locally advanced rectal cancer. However, radiation-related side effects could not be neglected. But this multimodality strategy failed to improve survival. Neoadjuvant chemotherapy alone may be an alternative strategy to minimize treatment-related toxicities without compromising the oncology outcome. Thus, patients with MRI-defined CRM-positive rectal cancer will receive 6 cycles of neoadjuvant treatment with FOLFOXIRI followed by surgery. The purpose of the study is to evaluate the efficacy of FOLFOXIRI alone as neoadjuvant treatment in treating patients with locally advanced rectal cancer.

DETAILED DESCRIPTION:
Preoperative chemoradiotherapy has been considered for years the standard treatment to patients with locally advanced rectal cancer. However, this multi-modality treatment has been questioned since more evidences suggested that radiotherapy may not be a necessary component of this treatment, and by omitting radiotherapy it have the advantage of reducing acute and late treatment-related toxicities. Given the high anti-tumor of systemic chemotherapy alone, any patients with CRM involvement could be theoretically deemed candidate for an approach in which radiotherapy is delivered preoperatively if a substantial tumor downsizing is not achieved after upfront systemic chemotherapy or postoperatively if the pathologic CRM is involved. This single phase Ⅱ trial was aimed to evaluate the efficacy of FOLFOXIRI in treating patients with MRI-defined CRM-positive rectal cancer. All patients will receive the regimen every 2 weeks for 3 cycles. MRI of the pelvic will be performed after 3 cycles of chemotherapy to assess clinical response. If the tumor responds after 3 cycles of treatment, the patient will continue for another 3 cycles of treatment before surgery under the decision of MDT. On the contrary, if the tumor shows no response, radiotherapy will be given before operation. After surgery and pathologic CRM is not involved, 6 cycles of mFOLFOX6 will be given as adjuvant chemotherapy, otherwise postoperative radiotherapy will be given if the pathologic CRM is involved.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adenocarcinoma of the rectum
* Age: 18-70years old
* Signed informed consent; able to comply with study and/or followup procedures
* Stage of the primary tumor may be determined by MRI as CRM positive
* Tumor amenable to curative resection
* Adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment:
* Leukocytes ≥ 3.0 x109/ L, absolute neutrophil count (ANC) ≥ 1.5 x109/ L, platelet count ≥ 100 x109/ L, hemoglobin (Hb) ≥ 9g/ dL.
* Total bilirubin ≤1.5 x the upper limit of normal (ULN).
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 x ULN.
* Alkaline phosphatase limit ≤ 5x ULN.
* Amylase and lipase ≤ 1.5 x the ULN.
* Serum creatinine ≤ 1.5 x the ULN.
* No renal disease that would preclude study treatment or followup
* ECOG status: 0～1

Exclusion Criteria:

* Hypersensitivity to fluorouracil, oxaliplatin or irinotecan.
* Less than 4 weeks since prior participation in any investigational drug study
* History of invasive rectal malignancy, regardless of disease free interval
* Uncontrolled hypertension
* Cardiovascular disease that would preclude study treatment or followup
* Lack of upper gastrointestinal tract integrity or malabsorption syndrome，active upper gastrointestinal tract bleeding
* Synchronous colon cancer
* Pregnant or nursing
* Other malignancy within the past 5 years except effectively treated squamous cell or basal cell skin cancer, melanoma in situ, carcinoma in situ of the cervix, or carcinoma in situ of the colon or rectum
* No psychiatric or addictive disorders, or other conditions that, in the opinion of the investigator, would preclude study participation
* patients refused to signed informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
The rate of negative circumferential margin status | 30 days
  Evaluation of the circumferential margin status (positive or negative) in the rectal specimen according international consensus (positive margin if tumor ≤ 1mm from circumferential margin)
The rate of R0 resection | 30 days
  Evaluation of the resection margin status (positive or negative) in the rectal specimen

SECONDARY OUTCOMES:
The rate of tumor downstaging to stage 0 and stage Ⅰ | 2 years
  Tumor downstaging from stage Ⅲ to pathologica complete response （stage 0） and stage Ⅰ
the local recurrence rate | 3 year
  the rate of patients with local recurrence within 3 years
Recurrence free survival | 3 year
  3 years recurrence free survival of this group of patients
Reported Adverse events | 3 years
  Number of patients with adverse events and severity according to NCI CTC 4.0 after treatment with this regimen

CONTACTS AND LOCATIONS:
Overall Officials: Yuzhou Qin, Study Director — Affiated Tumor Hospital of Guangxi Medical University
Locations (1):
- Affiliated Tumor Hospital of Guangxi Medical University, Nanning, Guangxi Autonomous Region, China

IPD SHARING:
Plan to Share IPD: No